CLINICAL TRIAL: NCT04170283
Title: An Open-label, Multi-center, Long-term Extension Study of Zanubrutinib (BGB-3111) Regimens in Patients With B-cell Malignancies
Brief Title: Long-term Extension Study of Zanubrutinib (BGB-3111) Regimens in Participants With B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-LTE1
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: B-cell Malignancies
Keywords: Zanubrutinib; Bruton's tyrosine kinase (BTK) inhibitor; long-term extension
MeSH Terms: interventions — zanubrutinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zanubrutinib (BGB-3111) (Experimental): All participants to receive open-label zanubrutinib
  Interventions: Drug: Zanubrutinib
- Zanubrutinib in combination with Tislelizumab (Experimental): Participants to receive the combination as in the parent study (Australia Only)
  Interventions: Drug: Zanubrutinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Zanubrutinib — Participants will receive zanubrutinib at a dose of 160 mg twice daily (for a total daily dose of 320 mg), or the last dose level received in the BeiGene parent study.
  Other Names: BGB-3111
Drug: Tislelizumab — Patients in Australia who participated in a parent study that involved combination therapy of zanubrutinib and tislelizumab will receive tislelizumab at a dose of 200mg every 3 weeks..
  Other Names: BGB-A317
  Arms: Zanubrutinib in combination with Tislelizumab

SUMMARY:
The purpose of this study is to evaluate the long-term safety of zanubrutinib regimens in participants with B-cell malignancies who participated in a BeiGene parent study for zanubrutinib.

ELIGIBILITY:
1. Currently participating or participated recently in a BeiGene parent study
2. Intent to continue or start zanubrutinib treatment after any of the following:

   1. At time of final analysis or study closure of the eligible BeiGene parent study
   2. At time of progressive disease (PD); and investigator, patient and medical monitor agree it is in the patient's best interest
   3. At an alternative timepoint for an alternative reason
3. Patient who is currently on zanubrutinib treatment:

   Does not meet any protocol-specified criteria for zanubrutinib hold or permanent discontinuation, and, in the opinion of the investigator, will continue to benefit from zanubrutinib treatment
4. Zanubrutinib-naive patient:

   Must meet the following criteria ≤ 15 days before first dose of study drug:
   1. Platelets ≥ 50,000/mm3
   2. Absolute neutrophil count ≥ 750/mm3
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal
   4. Serum total bilirubin ≤ 3 x upper limit of normal (not required for Gilbert Syndrome)
   5. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≤ 480 msec
   6. No known New York Heart Association (NYHA) Class III or IV congestive heart failure
   7. Creatinine clearance ≥ 30 mL/min
5. Female participants of childbearing potential and nonsterile males must be willing to use a highly effective method of birth control.

Key Exclusion Criteria:

1. Permanently discontinued from zanubrutinib treatment in the BeiGene parent study due to unacceptable toxicity, non-compliance with study procedures, or withdrawal of consent
2. Uncontrolled active systemic infection or recent infection requiring parenteral anti-microbial therapy
3. Life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of zanubrutinib, or put the study outcomes at undue risk
4. Concomitant chemotherapy, targeted therapy, radiation therapy, antibody-based therapies, or any prohibited concomitant therapy outlined in the protocol
5. Pregnant or lactating woman
6. Inability to comply with study procedures
7. Concurrent participation in another therapeutic clinical study
8. History of progressive disease (PD) while receiving a BTK inhibitor (excluding zanubrutinib)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 5 years
  Safety as assessed by incidence of all treatment-emergent adverse events (TEAEs) and serious AEs (SAEs)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) per investigator assessment | Up to 5 years
  Time from the starting date of zanubrutinib in the eligible BeiGene study to the date of first documentation of disease progression or death, whichever occurs first
Duration of Response (DOR) per investigator assessment | Up to 5 years
  Time from the date that response criteria are first met after the start of zanubrutinib in the eligible BeiGene study to the date that progressive disease (PD) is objectively documented or death, whichever occurs first
Overall Survival (OS) | Up to 5 years
  Time from the starting date of zanubrutinib in the eligible BeiGene study to the date of death due to any reason

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (152):
- United States (26):
  - Banner Md Anderson Cancer Center, Gilbert, Arizona
  - Carti Cancer Center, Little Rock, Arkansas
  - Rocky Mountain Cancer Centers Centennial, Centennial, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists Fort Myers, Fort Myers, Florida
  - Scri Florida Cancer Specialists North, St. Petersburg, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Forrest General Hospital Cancer Center, Hattiesburg, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Florham Park, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Clinical Research Alliance, Inc, Westbury, New York
  - Duke University Hospital, Durham, North Carolina
  - Oncology Associates of Oregon Willamette Valley Cancer Center, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Scri Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Fort Worth Cancer Center, Fort Worth, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Texas Oncology San Antonio Medical Center Usor, San Antonio, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc, Roanoke, Virginia
  - University of Washington Seattle Cancer Alliance, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
- Australia (26):
  - Paratus Clinical Research Woden, Canberra, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Border Medical Oncology, East Albury, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Brisbane Clinic For Lymphoma, Greenslopes, Queensland
  - John Flynn Private Hospital, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford PK, South Australia
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Barwon Health the Geelong Hospital, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- China (23):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Czechia (6):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Vseobecna Fakultni Nemocnice V Praze, Prague
  - University Hospital Vinohrady Hematology Department, Prague
- France (6):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Saint Louis, Paris
  - Chu Hopital Lyon Sud, PierreBenite
  - Chu Tours Hopital Bretonneau, Tours
- Srh Kliniken Landkreis Sigmaringen, Sigmaringen, Germany
- General Hospital of Athens Alexandra, Athens, Greece
- Italy (11):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Universita Degli Studi Di Modena Azienda Ospedaliere Policlinco, Modena
  - Aou Maggiore Della Carita, Novara
  - Irccs Policlinico San Matteo, Universita Degli Studi Di Pavi, Pavia
  - Unita Di Ematologia, Dipartimento Di Ematologia Ed Oncologia, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera S Maria Di Terni, Terni
  - Azienda Ospedaliera Citta Della Salute E Della Scienza Di Torino, Torino
  - Aou Santa Maria Della Misericordia Di Udine, Udine
- Japan (4):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kurume University Hospital, Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Aiiku Hospital, Sapporo, Hokkaido
- Netherlands (3):
  - Amsterdam Umc Amc, Amsterdam
  - Albert Schweitzer Ziekenhuis, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (7):
  - Auckland City Hospital, Auckland
  - Aotearoa Clinical Trials, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton Waikato
  - North Shore Hospital, Takapuna
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital (Ccdhb), Wellington
- Poland (9):
  - Interhem Opieka Szpitalna, Bialystok
  - Szpital Specjalist W Brzozowie,Podkarpacki Osrodek Onkologiczny, Brzozów
  - Szpital Uniwersytecki Nr Im Dr Jana Biziela, Bydgoszcz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Copernicus Podmiot Leczniczy Sp Z Oo Wojewodzkie Centrum Onkologii, Gdask
  - Malopolskie Centrum Medyczne Sc, Krakow
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Centrum Medyczne Pratia Poznan, Skorzewo Poznan
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan, Busan Gwang'yeogsi
  - Dong A University Hospital, Busan, Busan Gwang'yeogsi
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center Hematology Oncology, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall Dhebron, Barcelona
  - Ico Hug Trias I Pujol, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Ico Girona, Girona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Toledo, Toledo
- Sweden (2):
  - Skanes Universitetssjukhus I Lund, Lund
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Namik Kemal University, Tekirdağ, Turkey (Türkiye)
- United Kingdom (13):
  - Nhs Grampian Ppds, Aberdeen
  - Birmingham Heartlands Hospital, Birmingham
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - Kent and Canterbury Hospital, Canterbury
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie Hospital, Greater Manchester
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - St Jamess Institute of Oncology, Leeds
  - Barts Health Nhs Trust, London
  - University College Hospital, London
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Plymouth Hospitals Nhs Trust, Plymouth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Garcia-Sanz R, Owen RG, Jurczak W, Dimopoulos MA, McCarthy H, Cull G, Opat SS, Castillo JJ, Kersten MJ, Wahlin BE, Grosicki S, Prathikanti R, Tian T, Allewelt H, Cohen AC, Tam CS. Outcomes after transition from ibrutinib to zanubrutinib in patients with Waldenstrom macroglobulinemia from the ASPEN study. Blood Adv. 2025 Dec 23;9(24):6538-6546. doi: 10.1182/bloodadvances.2024015596. PMID 40924923
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198